CLINICAL TRIAL: NCT06020053
Title: Effect of Using Irrigations at Different Temperatures on Postoperative Period During the Extraction of Impacted Mandibular Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Ceren Dayanan, research assistant, Firat University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: FiratUniversitydentistry
Record Dates: First submitted 2023-07-20; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: irrigation,; third molar surgery,; temperature,

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One of the symmetrical Impacted Mandibular Third Molars, control group (No Intervention): Serum at room temperature (25°C) was applied to one of the mandibular impacted third molars
- One of the symmetrical Impacted Mandibular Third Molars, intervention group (Experimental): Serum at temperature (4°C) was applied to one of the mandibular impacted third molars
  Interventions: Procedure: saline irrigation at various temperatures (4°C, 25°C)

INTERVENTIONS:
Procedure: saline irrigation at various temperatures (4°C, 25°C) — cold serum application
  Arms: One of the symmetrical Impacted Mandibular Third Molars, intervention group

SUMMARY:
An Evaluation of the Effect of Using Irrigations at Different Temperatures on Pain, Edema, and Trismus During the Extraction of Bilateral Impacted Mandibular Third Molars: A Randomized Split-Mouth Clinical Trial

DETAILED DESCRIPTION:
Abstract Introduction: The surgical extraction of impacted wisdom teeth is a standard practice in dentistry. Unfortunately, inflammatory reactions such as discomfort, edema, and trismus frequently jeopardize patients' well-being after the extraction of third molars. Saline solutions at room temperature (25°C) are routinely used in impacted tooth extraction. Refrigerated serums were used to work with cold serum, and since the refrigerator temperature was 4°C, this study was designed to have a cold serum temperature of 4°C. This study aims to assess the influence of saline irrigation at various temperatures (4°C, 25°C) on postoperative edema, pain, and trismus after the extraction of impacted third molars.

Materials and Methods: Eighteen patients with bilateral symmetrical mandibular impacted third molars were enrolled in this split-mouth, randomized, prospective, double-blind clinical trial. For each patient, one side was irrigated with a solution at 4°C (test), and the other side was irrigated with a solution at room temperature (25°C) (control). Pain, trismus, and facial edema were noted on the 2nd, 4th, and 7th days. A Mann-Whitney U-test was used to compare pairs, and a Wilcoxon signed-rank test was used to compare groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 30 who were classified as ASA (American Society of Anesthesiologists)1 and who required the removal of impacted third molars on either the right or left side of the mandible;
* Presence of impacted mandibular third molars on panoramic radiographs, bilaterally symmetrical, with bone retention and bone removal for extraction, position B class 2 of impacted teeth according to the Pell and Gregory Classification System, and mesioangular position according to the Winter Classification;
* Absence of systemic disease and habitual smoking behavior and absence of an allergy to the drugs to be used postoperatively.

Exclusion Criteria:

* Patients with a history of taking antibiotics and analgesics for at least one month;
* Having an infection in the operation area and acute pericoronitis or severe periodontal disease before the operation;
* The existence of cysts and tumors within proximity of the impacted third molar.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Pain was noted on the 2nd, 4th, and 7th days. | on the 2nd, 4th, and 7th days.
  Pain was evaluated with a 10-unit visual analog scale (VAS), which was included in the patient follow-up form on the postoperative second, fourth, and seventh days.

SECONDARY OUTCOMES:
trismus was noted on the 2nd, 4th, and 7th days. | on the 2nd, 4th, and 7th days.
  For trismus, preoperative and postoperative mouth openings were evaluated on the second, fourth, and seventh days by measuring the maximum distance between the incisal surface of the right maxillary incisor and the incisal surface of the right mandibular incisor with a caliper.
facial edema was noted on the 2nd, 4th, and 7th days | on the 2nd, 4th, and 7th days.
  The level of facial edema was evaluated using Amin Laskin's protocol. Two measurements between four reference points were taken using a tape measure to assess facial edema. The distance between the tragus and the lip commissure and between the gonion and the lateral (outer) canthus of the eye were measured with a tape measure preoperatively and on the second, fourth, and seventh days after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: muhammet ozupek, Study Director — Firat University
Locations (1):
- Fırat Üniversitesi, Merkez, Elaziğ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No